CLINICAL TRIAL: NCT01429727
Title: The "Virtual" Multicenter Spontaneous Coronary Artery Dissection (SCAD) Registry
Acronym: SCAD
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Marysia Tweet, Principal Investigator, Mayo Clinic
Other Study IDs: 11-001852
Record Dates: First submitted 2011-08-30; First posted 2011-09-07 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Spontaneous Coronary Artery Dissection; SCAD
Keywords: Spontaneous coronary artery dissection; SCAD; coronary artery disease; myocardial infarction; coronary dissection
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous; Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SCAD Registry: Individuals who have experienced at least one episode of spontaneous coronary artery dissection.

SUMMARY:
The primary goal of this project is to describe the clinical and physiologic characteristics of Spontaneous Coronary Artery Dissections (SCAD) in order to increase awareness, understanding, treatment and prevention of a potentially fatal cardiovascular event.

This study will be a retrospective and prospective review of medical course and current health of men and women with SCAD.

DETAILED DESCRIPTION:
Spontaneous Coronary Artery Dissection (SCAD) is a relatively rare and poorly understood condition that has been reported to affect more women than men. The coronary arteries consist of three layers, and dissection occurs when two of these layers separate, enabling blood to flow into the space between the layers. As the blood accumulates, this can cause obstruction to normal blood flow within the heart, leading to chest pain, heart attack and even sudden death.

The medical community has much to learn about treatment and prevention of this potentially fatal cardiovascular event. Mayo Clinic is conducting two studies of SCAD. This study consists of building a database/registry of patients with SCAD (whether they have been patients at Mayo Clinic or not) to identify patterns of SCAD incidence, causes and associations that could guide future research. With participant consent, Mayo Clinic staff will request a copy of the original coronary angiogram when SCAD was diagnosed to confirm the diagnosis and determine eligibility. If eligible, study coordinators will contact the participant to provide more information about the studies and request a signed informed consent document.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been cared for at Mayo Clinic with a diagnosis of SCAD
* SCAD in women who are pregnant or within 12 months postpartum at the time of SCAD
* SCAD in individuals who self-identify as a member of a racial or ethnic group that is currently underrepresented in the registry. This would include anyone who identifies as: Black/African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, and any race with Hispanic ethnicity
* SCAD in a man
* SCAD in persons younger than 30 years of age
* SCAD within the past 2 weeks (acute)
* SCAD patient enrolling into any other Mayo Clinic SCAD Research Study
* SCAD in individuals who have a relative that has had a SCAD event

Persons with history of SCAD who are interested in participating in the study but do not meet the updated inclusion criteria will not be enrolled at this time. However, they will be given the option to share their contact information in order to be invited to future Mayo Clinic SCAD studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women with spontaneous coronary artery dissection (SCAD) as confirmed on angiogram.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2011-07; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Descriptive Data | Continuous time frame following index event for 2-10 years from study contact date.
  Obtain data regarding SCAD related risk factors, presenting characteristics, treatments and long term outcomes.

SECONDARY OUTCOMES:
Physical Health Update | Continuous time frame following index event for 2-10 years from study contact date.
  Record update on patient's current physical health and any relevant health events that may have occurred since the initial SCAD event.
Mental Health Update | Continuous time frame following index event for 2-10 years from study contact date.
  Record update on patient's current mental health status since the initial SCAD event.

CONTACTS AND LOCATIONS:
Overall Officials: Marysia S Tweet, M.D., M.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Tweet MS, Gulati R, Aase LA, Hayes SN. Spontaneous coronary artery dissection: a disease-specific, social networking community-initiated study. Mayo Clin Proc. 2011 Sep;86(9):845-50. doi: 10.4065/mcp.2011.0312. PMID 21878595
- [Background] Tweet MS, Hayes SN, Pitta SR, Simari RD, Lerman A, Lennon RJ, Gersh BJ, Khambatta S, Best PJ, Rihal CS, Gulati R. Clinical features, management, and prognosis of spontaneous coronary artery dissection. Circulation. 2012 Jul 31;126(5):579-88. doi: 10.1161/CIRCULATIONAHA.112.105718. Epub 2012 Jul 16. PMID 22800851
- [Background] Tweet MS, Gulati R, Williamson EE, Vrtiska TJ, Hayes SN. Multimodality Imaging for Spontaneous Coronary Artery Dissection in Women. JACC Cardiovasc Imaging. 2016 Apr;9(4):436-50. doi: 10.1016/j.jcmg.2016.01.009. PMID 27056163
- [Background] Krittanawong C, Tweet MS, Hayes SE, Bowman MJ, Gulati R, Squires RW, Hayes SN. Usefulness of Cardiac Rehabilitation After Spontaneous Coronary Artery Dissection. Am J Cardiol. 2016 May 15;117(10):1604-1609. doi: 10.1016/j.amjcard.2016.02.034. Epub 2016 Mar 2. PMID 27055757
- [Background] Henkin S, Negrotto SM, Tweet MS, Kirmani S, Deyle DR, Gulati R, Olson TM, Hayes SN. Spontaneous coronary artery dissection and its association with heritable connective tissue disorders. Heart. 2016 Jun 1;102(11):876-81. doi: 10.1136/heartjnl-2015-308645. Epub 2016 Feb 10. PMID 26864667
- [Background] Tweet MS, Gulati R, Hayes SN. What Clinicians Should Know Alphabout Spontaneous Coronary Artery Dissection. Mayo Clin Proc. 2015 Aug;90(8):1125-30. doi: 10.1016/j.mayocp.2015.05.010. PMID 26250728
- [Background] Prasad M, Tweet MS, Hayes SN, Leng S, Liang JJ, Eleid MF, Gulati R, Vrtiska TJ. Prevalence of extracoronary vascular abnormalities and fibromuscular dysplasia in patients with spontaneous coronary artery dissection. Am J Cardiol. 2015 Jun 15;115(12):1672-7. doi: 10.1016/j.amjcard.2015.03.011. Epub 2015 Mar 23. PMID 25929580
- [Background] Tweet MS, Hayes SN, Gulati R, Rose CH, Best PJ. Pregnancy after spontaneous coronary artery dissection: a case series. Ann Intern Med. 2015 Apr 21;162(8):598-600. doi: 10.7326/L14-0446. No abstract available. PMID 25894037
- [Background] Goel K, Tweet M, Olson TM, Maleszewski JJ, Gulati R, Hayes SN. Familial spontaneous coronary artery dissection: evidence for genetic susceptibility. JAMA Intern Med. 2015 May;175(5):821-6. doi: 10.1001/jamainternmed.2014.8307. PMID 25798899
- [Background] Silber TC, Tweet MS, Bowman MJ, Hayes SN, Squires RW. Cardiac rehabilitation after spontaneous coronary artery dissection. J Cardiopulm Rehabil Prev. 2015 Sep-Oct;35(5):328-33. doi: 10.1097/HCR.0000000000000111. PMID 25730096
- [Background] Eleid MF, Guddeti RR, Tweet MS, Lerman A, Singh M, Best PJ, Vrtiska TJ, Prasad M, Rihal CS, Hayes SN, Gulati R. Coronary artery tortuosity in spontaneous coronary artery dissection: angiographic characteristics and clinical implications. Circ Cardiovasc Interv. 2014 Oct;7(5):656-62. doi: 10.1161/CIRCINTERVENTIONS.114.001676. Epub 2014 Aug 19. PMID 25138034
- [Background] Hayes SN. Spontaneous coronary artery dissection (SCAD): new insights into this not-so-rare condition. Tex Heart Inst J. 2014 Jun 1;41(3):295-8. doi: 10.14503/THIJ-14-4089. eCollection 2014 Jun. No abstract available. PMID 24955045
- [Background] Liang JJ, Prasad M, Tweet MS, Hayes SN, Gulati R, Breen JF, Leng S, Vrtiska TJ. A novel application of CT angiography to detect extracoronary vascular abnormalities in patients with spontaneous coronary artery dissection. J Cardiovasc Comput Tomogr. 2014 May-Jun;8(3):189-97. doi: 10.1016/j.jcct.2014.02.001. Epub 2014 Apr 4. PMID 24939067
- [Background] Tweet MS, Gulati R, Hayes SN. Spontaneous Coronary Artery Dissection. Curr Cardiol Rep. 2016 Jul;18(7):60. doi: 10.1007/s11886-016-0737-6. PMID 27216840
- [Background] Lindor RA, Tweet MS, Goyal KA, Lohse CM, Gulati R, Hayes SN, Sadosty AT. Emergency Department Presentation of Patients with Spontaneous Coronary Artery Dissection. J Emerg Med. 2017 Mar;52(3):286-291. doi: 10.1016/j.jemermed.2016.09.005. Epub 2016 Oct 8. PMID 27727035
- [Background] Codsi E, Tweet MS, Rose CH, Arendt KW, Best PJM, Hayes SN. Spontaneous Coronary Artery Dissection in Pregnancy: What Every Obstetrician Should Know. Obstet Gynecol. 2016 Oct;128(4):731-738. doi: 10.1097/AOG.0000000000001630. PMID 27607875
- [Background] Eleid MF, Tweet MS, Young PM, Williamson E, Hayes SN, Gulati R. Spontaneous coronary artery dissection: challenges of coronary computed tomography angiography. Eur Heart J Acute Cardiovasc Care. 2018 Oct;7(7):609-613. doi: 10.1177/2048872616687098. Epub 2017 Jan 31. PMID 28139136
- [Background] Tweet MS, Codsi E, Best PJM, Gulati R, Rose CH, Hayes SN. Menstrual Chest Pain in Women With History of Spontaneous Coronary Artery Dissection. J Am Coll Cardiol. 2017 Oct 31;70(18):2308-2309. doi: 10.1016/j.jacc.2017.08.071. No abstract available. PMID 29073960
- [Background] Tweet MS, Hayes SN, Codsi E, Gulati R, Rose CH, Best PJM. Spontaneous Coronary Artery Dissection Associated With Pregnancy. J Am Coll Cardiol. 2017 Jul 25;70(4):426-435. doi: 10.1016/j.jacc.2017.05.055. PMID 28728686
- [Background] Tweet MS, Akhtar NJ, Hayes SN, Best PJ, Gulati R, Araoz PA. Spontaneous coronary artery dissection: Acute findings on coronary computed tomography angiography. Eur Heart J Acute Cardiovasc Care. 2019 Aug;8(5):467-475. doi: 10.1177/2048872617753799. Epub 2018 Jan 29. PMID 29376398
- [Background] Hayes SN, Kim ESH, Saw J, Adlam D, Arslanian-Engoren C, Economy KE, Ganesh SK, Gulati R, Lindsay ME, Mieres JH, Naderi S, Shah S, Thaler DE, Tweet MS, Wood MJ; American Heart Association Council on Peripheral Vascular Disease; Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Genomic and Precision Medicine; and Stroke Council. Spontaneous Coronary Artery Dissection: Current State of the Science: A Scientific Statement From the American Heart Association. Circulation. 2018 May 8;137(19):e523-e557. doi: 10.1161/CIR.0000000000000564. Epub 2018 Feb 22. PMID 29472380
- [Background] Waterbury TM, Tweet MS, Hayes SN, Prasad A, Lerman A, Gulati R. Coronary endothelial function and spontaneous coronary artery dissection. Eur Heart J Acute Cardiovasc Care. 2020 Feb;9(1):90-95. doi: 10.1177/2048872618795255. Epub 2018 Aug 20. PMID 30124050
- [Background] Tan NY, Hayes SN, Young PM, Gulati R, Tweet MS. Usefulness of Cardiac Magnetic Resonance Imaging in Patients With Acute Spontaneous Coronary Artery Dissection. Am J Cardiol. 2018 Nov 15;122(10):1624-1629. doi: 10.1016/j.amjcard.2018.07.043. Epub 2018 Aug 20. PMID 30220414
- [Background] Waterbury TM, Tweet MS, Hayes SN, Eleid MF, Bell MR, Lerman A, Singh M, Best PJM, Lewis BR, Rihal CS, Gersh BJ, Gulati R. Early Natural History of Spontaneous Coronary Artery Dissection. Circ Cardiovasc Interv. 2018 Sep;11(9):e006772. doi: 10.1161/CIRCINTERVENTIONS.118.006772. PMID 30354594
- [Background] Kok SN, Hayes SN, Cutrer FM, Raphael CE, Gulati R, Best PJM, Tweet MS. Prevalence and Clinical Factors of Migraine in Patients With Spontaneous Coronary Artery Dissection. J Am Heart Assoc. 2018 Dec 18;7(24):e010140. doi: 10.1161/JAHA.118.010140. PMID 30561271
- [Background] Adlam D, Olson TM, Combaret N, Kovacic JC, Iismaa SE, Al-Hussaini A, O'Byrne MM, Bouajila S, Georges A, Mishra K, Braund PS, d'Escamard V, Huang S, Margaritis M, Nelson CP, de Andrade M, Kadian-Dodov D, Welch CA, Mazurkiewicz S, Jeunemaitre X; DISCO Consortium; Wong CMY, Giannoulatou E, Sweeting M, Muller D, Wood A, McGrath-Cadell L, Fatkin D, Dunwoodie SL, Harvey R, Holloway C, Empana JP, Jouven X; CARDIoGRAMPlusC4D Study Group; Olin JW, Gulati R, Tweet MS, Hayes SN, Samani NJ, Graham RM, Motreff P, Bouatia-Naji N. Association of the PHACTR1/EDN1 Genetic Locus With Spontaneous Coronary Artery Dissection. J Am Coll Cardiol. 2019 Jan 8;73(1):58-66. doi: 10.1016/j.jacc.2018.09.085. PMID 30621952
- [Background] Turley TN, Theis JL, Sundsbak RS, Evans JM, O'Byrne MM, Gulati R, Tweet MS, Hayes SN, Olson TM. Rare Missense Variants in TLN1 Are Associated With Familial and Sporadic Spontaneous Coronary Artery Dissection. Circ Genom Precis Med. 2019 Apr;12(4):e002437. doi: 10.1161/CIRCGEN.118.002437. Epub 2019 Mar 19. PMID 30888838
- [Background] Johnson AK, Hayes SN, Sawchuk C, Johnson MP, Best PJ, Gulati R, Tweet MS. Analysis of Posttraumatic Stress Disorder, Depression, Anxiety, and Resiliency Within the Unique Population of Spontaneous Coronary Artery Dissection Survivors. J Am Heart Assoc. 2020 May 5;9(9):e014372. doi: 10.1161/JAHA.119.014372. Epub 2020 Apr 28. PMID 32342736
- [Background] Turley TN, O'Byrne MM, Kosel ML, de Andrade M, Gulati R, Hayes SN, Tweet MS, Olson TM. Identification of Susceptibility Loci for Spontaneous Coronary Artery Dissection. JAMA Cardiol. 2020 Aug 1;5(8):929-938. doi: 10.1001/jamacardio.2020.0872. PMID 32374345
- [Background] Hayes SN, Tweet MS, Adlam D, Kim ESH, Gulati R, Price JE, Rose CH. Spontaneous Coronary Artery Dissection: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Aug 25;76(8):961-984. doi: 10.1016/j.jacc.2020.05.084. PMID 32819471
- [Background] Tweet MS, Young KA, Best PJM, Hyun M, Gulati R, Rose CH, Hayes SN. Association of Pregnancy With Recurrence of Spontaneous Coronary Artery Dissection Among Women With Prior Coronary Artery Dissection. JAMA Netw Open. 2020 Sep 1;3(9):e2018170. doi: 10.1001/jamanetworkopen.2020.18170. PMID 32965500
- [Background] Kronzer VL, Tarabochia AD, Lobo Romero AS, Tan NY, O'Byrne TJ, Crowson CS, Turley TN, Myasoedova E, Davis JM 3rd, Raphael CE, Gulati R, Hayes SN, Tweet MS. Lack of Association of Spontaneous Coronary Artery Dissection With Autoimmune Disease. J Am Coll Cardiol. 2020 Nov 10;76(19):2226-2234. doi: 10.1016/j.jacc.2020.09.533. PMID 33153582
- [Background] Benson JC, Lehman VT, Verdoorn JT, Shlapak DP, Hayes SN, Tweet MS. Prevalence of Cervical Artery Abnormalities on CTA in Patients with Spontaneous Coronary Artery Dissection: Fibromuscular Dysplasia, Dissection, Aneurysm, and Tortuosity. AJNR Am J Neuroradiol. 2021 Aug;42(8):1497-1502. doi: 10.3174/ajnr.A7151. Epub 2021 May 13. PMID 33985951
- [Background] Turley TN, Kosel ML, Bamlet WR, Gulati R, Hayes SN, Tweet MS, Olson TM. Susceptibility Locus for Pregnancy-Associated Spontaneous Coronary Artery Dissection. Circ Genom Precis Med. 2021 Aug;14(4):e003398. doi: 10.1161/CIRCGEN.121.003398. Epub 2021 Aug 13. No abstract available. PMID 34384238
- [Background] Adlam D, Tweet MS, Gulati R, Kotecha D, Rao P, Moss AJ, Hayes SN. Spontaneous Coronary Artery Dissection: Pitfalls of Angiographic Diagnosis and an Approach to Ambiguous Cases. JACC Cardiovasc Interv. 2021 Aug 23;14(16):1743-1756. doi: 10.1016/j.jcin.2021.06.027. PMID 34412792
- [Background] Johnson AK, Tweet MS, Rouleau SG, Sadosty AT, Hayes SN, Raukar NP. The presentation of spontaneous coronary artery dissection in the emergency department: Signs and symptoms in an unsuspecting population. Acad Emerg Med. 2022 Apr;29(4):423-428. doi: 10.1111/acem.14426. Epub 2021 Dec 26. PMID 34897898
- [Background] Tarabochia AD, Tan NY, Lewis BR, Slusser JP, Hayes SN, Best PJM, Gulati R, Deshmukh AJ, Tweet MS. Association of Spontaneous Coronary Artery Dissection With Atrial Arrhythmias. Am J Cardiol. 2023 Jan 1;186:203-208. doi: 10.1016/j.amjcard.2022.09.032. Epub 2022 Oct 31. PMID 36328832
- See also: Information for patients about spontaneous coronary artery dissection — http://www.mayoclinic.org/spontaneous-coronary-artery-dissection/
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials